CLINICAL TRIAL: NCT04082000
Title: A Phase 2a Study Examining the Safety and Efficacy of BOL-DP-o-04 Sublingual Drops for Treating Diabetic Neuropathy
Brief Title: Phase 2a Study Examining the Safety and Efficacy of BOL-DP-o-04 for Treating Diabetic Neuropathy
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: study stopped due to company strategic prioritization
Sponsor: Breath of Life International Pharma Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BOL-P-4
Record Dates: First submitted 2019-08-31; First posted 2019-09-09 (Actual); Last update posted 2021-03-24 (Actual); Status verified 2021-03

CONDITIONS: Diabetic Neuropathy
MeSH Terms: conditions — Diabetic Neuropathies

STUDY DESIGN:
Intervention Model Description: Double-blind
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Triple (Participant, Investigator, Outcomes Assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BOL-DP-o-04 (Experimental)
  Interventions: Drug: BOL-DP-o-04
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BOL-DP-o-04 — BOL-DP-o-04
  Arms: BOL-DP-o-04
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled Phase 2a Study Examining the Safety and Efficacy of BOL-DP-o-04 for Treating Diabetic Neuropathy

DETAILED DESCRIPTION:
A Phase 2a, two-center, randomized, double-blind, placebo-controlled study in which subjects will be randomized to receive either BOL-DP-o-04 or placebo in addition to Standart of Care. The study evaluates the effect of BOL-DP-o-04 for Diabetic Neuropathy. The study includes a screening period up to three weeks followed by a 12-week treatment period

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects with Type 1 or Type 2 diabetes
2. Diabetes duration of at least 1 year
3. HbA1c 6%-12%
4. 18 years of age or older
5. Diabetic neuropathy for at least 6 months
6. Failed or uncontrolled treatment of diabetic neuropathy following treatment with at least two drugs from the following drug list (Pregabalin / Dulexatine/ Amitriptyline / gabapentin /carbamazepine) for a duration of at least three months for each drug
7. Score equal or above 50% in DN4 questionnaire

Exclusion Criteria:

1. Neuropathic pain other than diabetic
2. A score of less than 50% on DN4 questionnaire
3. History of substance abuse (alcohol / illegal drugs)
4. History of cannabis or cannabis product usage in the last three months
5. Any decompensated chronic disease
6. Pregnancy/lactation
7. Participant in other clinical trial during the last 30 days
8. A current of history of cancer during the last year
9. Any mental/psychiatric illness in first-degree relative in a young patient <30 years old.
10. Any food allergy
11. History of amputation
12. Any disorder which in the investigator's opinion might jeopardize the subject's safety or compliance with the protocol
13. Patients with known allergy to one or more of the study drug components.
14. Patient with uncontrolled congestive heart failure
15. Subjects who get the following medications: opiates, Primidone, Phenobarbitol, carbamazepine, Rifampicin, Rifabutin, Troglitazone, and Hypericum perforatum
16. Patients with psychotic state in the past or anxiety disorder
17. Subject with a history of addiction or drug abuse.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2020-11-04 (Actual); Study Completion 2020-11-04 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with >30% reduction in neuropathic pain | Baseline to week 15
  Assessed by the DN4 questionnaire
Adverse Events (AEs) and Serious Adverse Events (SAEs) | First treatment upto 15 weeks
  All AEs will be recorded, whether considered minor or serious, drug-related or not

SECONDARY OUTCOMES:
Improvement of QoL from baseline | Baseline to 15 weeks
  Assessed by Diabetes Quality of Life Questionnaire (DQOL) questionnaire
Change in HbA1c | Baseline to 15 weeks
  Assessed by HbA1c blood levels
Percentage of patients achieving HbA1c < 7% | Baseline to 15 weeks
  Assessed by HbA1c blood levels
Change from baseline of blood pressure | Baseline to 15 weeks
  blood pressure measurement
Change in weight | Baseline to 15 weeks
  weight measured by Kg
Improvement in sleep disturbance | Baseline to 15 weeks
  Assessed by the sleep disturbance (PSQI) questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Wolfson Medical Center, Holon, Israel